CLINICAL TRIAL: NCT01969864
Title: College and University Student Intervention to Increase Consent for Organ Donation
Brief Title: University Student Intervention to Increase Organ Donation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, John Daryl Thornton, MD, MPH, Associate Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: P60MD00265DT3; 1P60MD002265-01 (NIH)
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Organ Donation; Health Behavior
Keywords: Randomized Controlled Trial; Healthcare Disparities
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- HRSA Video Intervention (Experimental): 5-minute video on organ donation from U.S. Department of Health and Human Services
  Interventions: Behavioral: HRSA Video Intervention
- PI Video Intervention (Experimental): 5-minute video on organ donation created in part by the principal investigator.
  Interventions: Behavioral: PI Video Intervention
- CDC Health Website Intervention (Placebo Comparator): This control intervention will include text from the CDC website on health and wellness.
  Interventions: Behavioral: CDC Health Website Intervention

INTERVENTIONS:
Behavioral: HRSA Video Intervention
  Arms: HRSA Video Intervention
Behavioral: PI Video Intervention
  Arms: PI Video Intervention
Behavioral: CDC Health Website Intervention
  Arms: CDC Health Website Intervention

SUMMARY:
The purpose of this study is to determine the effect of brief organ donation video interventions on consent for organ donation among college and university students. Our hypothesis is that the organ donation video interventions will be superior to lay health websites for increasing organ donation consent.

DETAILED DESCRIPTION:
This randomized controlled trial will involve 600 intervention and 600 control university students. Students will be randomized to 1 of 3 arms: a 5-minute video by the U.S. Department of Health and Human Services, a 5-minute video by the study principal investigator, or a health-related website by the Centers for Disease Control. After viewing the intervention, participants will be asked questions including whether they would like to consent to organ donation on their state electronic registry.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled student
* English speaking
* No severe visual or auditory impairment
* Citizen of the United States of America
* Not a currently registered organ donor
* Has a driver's license, state identification card, or learner's permit from one of the 50 states

Exclusion Criteria:

* Not a currently enrolled student
* Limited English proficiency
* Severe visual or auditory impairment
* Registered organ donor
* Does not have an active driver's license, state identification card, or learner's permit from one of the 50 states

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2261 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Proportion of students who agreed to consent to donation on the state electronic donor registry | One day
  Proportion of students who agreed to consent to donation on the state electronic donor registry

SECONDARY OUTCOMES:
Proportion of students who were willing to donate within 6 months | One day
  Proportion of students who were willing to donate within 6 months
Intervention quality | One day
  Student-reported quality of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: John D Thornton, MD, MPH, Principal Investigator — Case Western Reserve University
Locations (3):
- United States (3):
  - Baldwin Wallace University, Berea, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland State University, Cleveland, Ohio

REFERENCES:
- [Derived] Thornton JD, Patrick B, Sullivan C, Albert JM, Wong KA, Allen MD, Kimble L, Mekesa H, Bowen G, Sehgal AR. Comparing web-based video interventions to enhance university student willingness to donate organs: A randomized controlled trial. Clin Transplant. 2019 Apr;33(4):e13506. doi: 10.1111/ctr.13506. Epub 2019 Mar 13. PMID 30793375